CLINICAL TRIAL: NCT04261998
Title: The Effects of Sevice-learning in Physiotherapy Students: Exercise Program for Patients With Heart Transplantation and Acute Coronary Syndrome
Brief Title: Sevice-learning in Physiotherapy and Heart Transplantation and Acute Coronary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Elena Marques-Sule, Doctor in Physiotherapy, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H1542195894247
Record Dates: First submitted 2019-01-02; First posted 2020-02-10 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Heart Transplantation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Service-learning group (Experimental): Intervention group will perform a service-learning program with real patients with heart transplantation and coronary syndrome, and will have to perform a physical therapy program adapted to a real patient. Two meetings will be performed in order to establish groups, explain the project and search information based on evidence in scientific databases. In addition, three meetings with patients will be stated in order to establish the adapted program based on the real patient's needs and characteristics.
  Interventions: Other: Service-learning program
- Control group (No Intervention): Control group will perform a physical therapy program for heart transplantation and coronary syndrome, but without meeting real patients. One meeting will be performed in order to establish groups and search information based on evidence in scientific databases.

INTERVENTIONS:
Other: Service-learning program — Intervention group will perform a service-learning program with real patients with heart transplantation, and will have to perform a physical therapy program adapted to a real patient. Two meetings will be performed in order to establish groups, explain the project and search information based on evidence in scientific databases. In addition, three meetings with patients will be stated in order to establish the adapted program based on the real patient's needs and characteristics.
  Arms: Service-learning group

SUMMARY:
A service-learning programme in physiotherapy students will be performed. 30 physiotherapy students will be randomly assigned to an intervention group (n=16) or to a control group (n=16). Intervention group will perform a service-learning program with real patients with heart transplantation, and will have to perform a physical therapy program adapted to a real patient. Two meetings will be performed in order to establish groups, explain the project and search information based on evidence in scientific databases. In addition, three meetings with patients will be stated in order to establish the adapted program based on the real patient's needs and characteristics. The control group will have to perform a physiotherapy program without meeting real patients.

DETAILED DESCRIPTION:
This study aims at determining the effect of a Service-Learning program on knowledge, ethical sensitivity and acquired transversal competences. On the other hand, we aim at evaluating the service performed, the skills acquired, the participation, the degree of participatory evaluation and the level of satisfaction of the intervention group. All variables will be measured with validated scales or questionnaires.

Both groups will have to describe the specific characteristics of the program, different phases of the process, types of exercises recommended, contraindications, safety ranges with respect to the intensity of the exercise, ways of calculating the intensity and self-control. Likewise, they will have to defend the usefulness and duration of the final product through an oral presentation of the program to the patients themselves. Finally, the possible doubts that should exist will be solved.

ELIGIBILITY:
Inclusion Criteria:

* Physiotherapy students

Exclusion Criteria:

* Prior courses on cardiac rehabilitation

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Ethical sensitivity | baseline
  Ethical sensitivity Questionnaire, composed of of 9 items with six possible responses (Likert scale from 1, indicating total disagreement, to 6, indicating total agreement). The minimum score is 9 and the maximum score is 54. The more score, the more ethical sensitivity. Cronbach's alpha=0.76
Ethical sensitivity | 3 months
  Ethical sensitivity Questionnaire, composed of of 9 items with six possible responses (Likert scale from 1, indicating total disagreement, to 6, indicating total agreement). The minimum score is 9 and the maximum score is 54. The more score, the more ethical sensitivity. Cronbach's alpha=0.76

SECONDARY OUTCOMES:
Service performed (by the students of the experimental group) | 3 months
  Service-learning Questionnaire, using the part of the questionnaire about service
Skills acquired (by the students of the experimental group) | 3 months
  Service-learning Questionnaire, using the part of the questionnaire about skills
Participation (of the students of the experimental group) | 3 months
  Service-learning Questionnaire,using the part of the questionnaire about participation
Degree of participatory evaluation (of the students of the experimental group) | 3 months
  Questionnaire of Participatory evaluation, Service-learning and university
Level of satisfaction (of the students of the experimental group) | 3 months
  ad-hoc satisfaction questionnaire
Knowledge on physiotherapy in heart transplantation | baseline
  A 10-question test exam will be created ad-hoc
Knowledge on physiotherapy in heart transplantation | 3 months
  A 10-question test exam will be created ad-hoc
Acquired transversal competences | baseline
  Questionnaire of Higher education, transversal skills and gender, consisted of 6 items about gender and competencies (Likert scale of 7 points: level 4 was set as neutral, scores above 4 were considered positive, and those below 4 were taken as negative scores)
Acquired transversal competences | 3 months
  Questionnaire of Higher education, transversal skills and gender, consisted of 6 items about gender and competencies (Likert scale of 7 points: level 4 was set as neutral, scores above 4 were considered positive, and those below 4 were taken as negative scores)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Marques-Sule, PT, PhD, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain